CLINICAL TRIAL: NCT02041208
Title: A Retrospective, Observational Study to Evaluate Hemoglobin Variability in Kidney Transplant Recipients With Chronic Renal Anemia.
Brief Title: Variability of Hemoglobin Levels After Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Sociedad Española de Trasplante (Other)
Responsible Party: Sponsor
Other Study IDs: SET-ANE-2011-01
Record Dates: First submitted 2013-12-19; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Renal Anemia
Keywords: Chronic renal anemia; Hemoglobin; Kidney transplant
MeSH Terms: interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: kidney transplantation — kidney transplantation

SUMMARY:
The purpose of this study es to determine hemoglobin variability in kidney transplant recipients with chronic renal anemia.

DETAILED DESCRIPTION:
The primary endpoint of the study is hemoglobin level variability. For determination of this variability, the following patterns of hemoglobin level change will be established:

* Target range hemoglobin (TRH): patients with hemoglobin values in the range of 11.0-12.0g/dl throughout the study period.
* Low hemoglobin (LH): patients with levels below 11.0g/dl
* High hemoglobin (HH): patients with levels above 12.0g/dl
* Low-amplitude fluctuation with low hemoglobin (LALH): patients with at least one measurement of hemoglobin levels <11.0g/dl and at least one measurement in the range of 11.0-12.0g/dl, but without hemoglobin measurements >12.0g/dl.
* Low-amplitude fluctuation with high hemoglobin (LAHH): patients with at least one measurement of hemoglobin levels >12.0g/dl and at least one measurement in the range of 11.0-12.0g/dl, but without hemoglobin measurements <11.0g/dl.
* High-amplitude fluctuation (HAH): patients with at least one measurement of hemoglobin levels <11.0g/dl and at least one measurement >12.0g/dl.

Secondary objectives:

* To determine potential factors influencing hemoglobin variability.
* To assess the influence of hemoglobin variability on cardiovascular risk of patients according to the REGICOR function at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > or = 18 years.
* Kidney transplant recipients with chronic renal failure stage 3 (glomerular filtration rate: 30-59ml/min/1.73m2), 4 (glomerular filtration rate: 15-29ml/min/1.73m2) or 5 (glomerular filtration rate: <15ml/min/1.73m2) at the start of the study follow-up period.
* Diagnosis of anemia and drug treatment initiated or changed subsequent to June 29, 2010 (date on which the latest recommendation by European Renal Best Practice on the target range for hemoglobin levels were published)
* Patients capable of giving their informed consent to participate in the study and who agree to participate by signing the informed consent form.

Exclusion Criteria:

* Patients whose medical history lacks measurements of hemoglobin levels every three months (±1 month) during the year of study follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult kidney transplant recipients with chronic renal anemia.
Sampling Method: Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is hemoglobin level variability | the study includes the retrospective collection of information from the medical records of patients over a period of one year.
  For determination of this variability, the following patterns of hemoglobin level change will be established:
  * Target range hemoglobin (TRH): patients who maintain hemoglobin values in the range of 11.0-12.0g/dl throughout the study period. - Low hemoglobin (LH): patients with hemoglobin levels below 11.0g/dl.
  * High hemoglobin (HH): patients with hemoglobin levels above 12.0g/dl.
  * Low-amplitude fluctuation with low hemoglobin (LALH): patients with at least one measurement of hemoglobin levels <11.0g/dl and at least one measurement in the range of 11.0-12.0g/dl, but without hemoglobin measurements >12.0g/dl.
  * Low-amplitude fluctuation with high hemoglobin (LAHH): patients with at least one measurement of hemoglobin levels >12.0g/dl and at least one measurement in the range of 11.0-12.0g/dl, but without hemoglobin measurements <11.0g/dl.
  * High-amplitude fluctuation (HAH): patients with at least one measure of hemoglobin levels <11.0g/dl and at least one measurement >12.0g/dl

SECONDARY OUTCOMES:
Estimation of cardiovascular risk of patients | at the end of the study period (one year after the start of data recording)
  according to the REGICOR function (acronym Girona Heart Registry)
Potential factors influencing hemoglobin variability | Both baseline data and the changes recorded on the visit at month 12 will be considered.
  Demographic and anthropometric data, comorbidities, concomitant medication, and data on transplant, chronic renal failure, renal anemia treatment and possible hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Sánchez Fructuoso, Coordinator, Study Chair — Hospital San Carlos, Madrid; Domingo Hernández, Md, Principal Investigator — Hospital Carlos Haya de Málaga; Teresa García, Md, Principal Investigator — Hospital Universitario Puerta del Mar; Ernesto Gómez Huertas, Md, Principal Investigator — Hospital Univ. Central de Asturias; Francisco Llamas Fuentes, Md, Principal Investigator — Complejo Hospitalario Univ. de Albacete; Juan Carlos Ruiz San Millán, Coordinator, Study Chair — Hospital Uni. Marqués de Valdecilla; Luis Guirado Perich, Coordinator, Study Chair — Fundación Puigvert; José Vicente Torregrosa, Md, Principal Investigator — Hospital Clinic of Barcelona; Francesc Moreso, Md, Principal Investigator — Hospital Univ. Vall d´Hebron; Ricardo Lauzurica Valdemoros, Md, Principal Investigator — Hospital Univ. Germans Trias i Pujol; María Luisa Mir Fontana, Md, Principal Investigator — Hospital del Mar; Alberto Martínez Castelao, Md, Principal Investigator — Hospital Univ. de Bellvitge; Rafael Romero Burgos, Md, Principal Investigator — Complejo Hospitalario Univ. de Santiago; Gonzalo Gómez, Md, Principal Investigator — Hospital Son Espases; Roberto Gallego Samper, Md, Principal Investigator — Hospital Univ. Dr. Negrín; Esther González Monte, Md, Principal Investigator — Hospital 12 de Octubre; Carlos Jiménez Martín, Md, Principal Investigator — Hospital Univ. La Paz; Manuel Rengel Aranda, Md, Principal Investigator — Hospital Univ. Gregorio Marañón; Carmen Bernis, Md., Principal Investigator — Hospital Univ. La Princesa; Pedro Errasti Goenaga, Md., Principal Investigator — Clínica Univ. de Navarra; Jaime Sánchez Plumed, Md, Principal Investigator — Hospital Univ. La Fe; Antonio Franco Esteve, Md, Principal Investigator — Hospital General Universitario de Alicante
Locations (22):
- Spain (22):
  - Complejo Hospitalario Universitario de Albacete, Albacete, Albacete
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Fundación Puigvert, Barcelona, Barcelona
  - Hospital Universitario Vall d´Hebron, Barcelona, Barcelona
  - Hospital Clinic i Provincial, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Hospital Universitario Dr. Negrín, Gran Canaria, Gran Canaria
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Universitario la Princesa, Madrid, Madrid
  - Hospital UniversitarioGregorio Marañón, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Carlos Haya de Málaga, Málaga, Málaga
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario La Fe, Valencia, Valencia